CLINICAL TRIAL: NCT00077207
Title: A Pilot Study Using Carboplatin, Vincristine And Temozolomide For Children ≤ 10 Years With Progressive/Symptomatic Low-Grade Gliomas
Brief Title: Carboplatin, Vincristine, and Temozolomide in Treating Children With Progressive and/or Symptomatic Low-Grade Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0223; CDR0000350005 (Other: Clinical Trials.gov); COG-ACNS0223 (Other: Children's Oncology Group); NCI-2012-02572 (Other: NCI)
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Brain Tumor; Central Nervous System Tumor
Keywords: untreated childhood cerebellar astrocytoma; untreated childhood visual pathway and hypothalamic glioma; childhood spinal cord neoplasm; childhood oligodendroglioma; childhood low-grade cerebral astrocytoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Spinal Cord Neoplasms; Oligodendroglioma | interventions — Carboplatin; Temozolomide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carboplatin, vincristine sulfate, temozolomide) (Experimental): Induction therapy: Patients receive carboplatin IV (175/m2) over 1 hour on days 1, 8, 15, and 22; vincristine IV (1.5 mg/m2) on days 1, 8, 15, 22, 29, and 36; and oral temozolomide (200 mg/m2) on days 43-47. Four weeks after the completion of induction therapy, patients achieving stable or responding disease proceed to maintenance therapy. Maintenance therapy: Patients receive carboplatin (175/m2) and temozolomide (200 mg/m2) as in induction therapy and vincristine IV ((1.5 mg/m2) day 1 of weeks 10,11,12. Treatment repeats every 10 weeks for a total of 6 courses in the absence of disease progression.
  Interventions: Drug: carboplatin; Drug: temozolomide; Drug: vincristine sulfate

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Paraplatin; NSC #241240
Drug: temozolomide — Given orally
  Other Names: Temodar; NSC# 362856
Drug: vincristine sulfate — Given IV
  Other Names: Oncovin; VCR; LCR; NSC #67574

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, vincristine, and temozolomide, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: This pilot study is studying giving carboplatin and vincristine together with temozolomide in treating children with progressive and/or symptomatic low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and toxicity of an induction and maintenance regimen comprising carboplatin, vincristine, and temozolomide in children with progressive and/or symptomatic low-grade gliomas.

Secondary

* Determine response rate in patients treated with this regimen.
* Determine 3-year progression-free survival and overall survival of patients treated with this regimen.
* Correlate response and progression-free survival with the genomic profile of tumors in patients treated with this regimen.

OUTLINE: This is a pilot study.

* Induction therapy: Patients receive carboplatin IV over 1 hour on days 1, 8, 15, and 22; vincristine IV on days 1, 8, 15, 22, 29, and 36; and oral temozolomide on days 43-47. Four weeks after the completion of induction therapy, patients achieving stable or responding disease proceed to maintenance therapy.
* Maintenance therapy: Patients receive carboplatin and temozolomide as in induction therapy and vincristine IV on days 1, 8, and 15. Treatment repeats every 10 weeks for a total of 6 courses in the absence of disease progression.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 30-50 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed progressive and/or symptomatic low-grade glioma, including any of the following:

  * WHO grade I or II astrocytoma
  * Grade I or II oligodendrogliomas
  * Mixed oligodendrogliomas
  * Gangliogliomas
* Measurable disease
* Progressive and/or symptomatic supratentorial or spinal cord tumors that cannot be removed for anatomical reasons are allowed
* Optic pathway tumors allowed provided there is evidence of progressive disease by MRI and/or symptoms of deteriorating vision, progressive hypothalamic/pituitary dysfunction, or diencephalic syndrome
* Dorsally exophytic brainstem gliomas that were previously resected more than 50% are allowed provided the residual tumor shows progression (with or without symptoms)
* No diffuse brain stem tumors
* No type 1 neurofibromatosis

PATIENT CHARACTERISTICS:

Age

* 10 and under

Performance status

* ECOG 0-2
* Lansky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 8.0 gm/dL
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 2.5 times ULN

Renal

* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR
* Creatinine ≤ 0.8 mg/dL (age 5 and under) OR ≤ 1.0 mg/dL (age 6 to10)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunomodulating agents

Chemotherapy

* No other concurrent anticancer chemotherapy

Endocrine therapy

* Prior corticosteroids allowed
* No concurrent corticosteroids except for the treatment of increased intracranial pressure

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* Prior surgery allowed

Other

* No other prior therapy

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2004-07; Primary Completion 2010-03 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murali M. Chintagumpala, MD, Study Chair — Texas Children's Cancer Center
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Chintagumpala MM, Adesina A, Morriss MC, et al.: A pilot study using carboplatin, vincristine, and temozolomide for children with progressive/symptomatic low-grade glioma: A Children's Oncology Group (COG) study. [Abstract] J Clin Oncol 28 (Suppl 15): A-9539, 2010.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Carboplatin, Vincristine Sulfate, Temozolomide)
Started | 66
Completed | 36
Not Completed | 30
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 12
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 6
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Carboplatin, Vincristine Sulfate, Temozolomide)
Number analyzed (Participants) | 66
Age, Continuous [Median (Full Range); unit: years] | 4 [0 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 49
  More than one race | 0
  Unknown or Not Reported | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 61
  Canada | 1
  Australia | 4

OUTCOME MEASURES:

1. Primary Outcome: Short Term Feasibility Success
Description: Success is defined as the completion of induction plus one cycle of maintenance within 24 weeks of enrollment without more than a 25% reduction in either carboplatin or temozolomide dosage.
  Failure to complete the induction and one cycle of maintenance within 24 weeks counts as a short-term-feasibility failure.
Time Frame: 24 weeks
Population: Fourteen (14) patients were considered not evaluable for short-term toxicity because: ineligible - 1 patient; progression during induction - 9 patients; progression during maintenance 2 patients; parent preference - 1 patient and infection resulting in termination of protocol therapy - 1 patient.
Measure: Number; unit: participants
Arm/Group | Treatment (Carboplatin, Vincristine Sulfate, Temozolomide)
Number analyzed (Participants) | 52
participants | 25

2. Primary Outcome: Long Term Feasibility Success
Description: Success is defined as the completion of induction plus four cycles of maintenance within 60 weeks of enrollment without more than a 25% reduction in either carboplatin or temozolomide dosage.
  If the participant completes all therapy within 60 weeks the patient is a long-term feasibility success. As such, a patient who experiences short term feasibility failure can be classified as a long-term feasibility success.
Time Frame: 60 weeks
Population: Fourteen (14) patients were considered not evaluable for long-term toxicity because: ineligible - 1 patient; progression during induction - 9 patients; progression during maintenance 2 patients; parent preference - 1 patient and infection resulting in termination of protocol therapy - 1 patient.
Measure: Number; unit: participants
Arm/Group | Treatment (Carboplatin, Vincristine Sulfate, Temozolomide)
Number analyzed (Participants) | 52
participants | 41

3. Secondary Outcome: Number of Participants Who Experienced Toxic Death
Description: Primary safety endpoints are (1) the occurrence of toxic death, which is death during treatment that is not primarily attributable to disease progression, and (2) the occurrence of grade 4 allergy to carboplatin.
Time Frame: Up to 6 years after the start of protocol therapy
Population: Sixty-five (65) eligible patients were enrolled and received protocol therapy. These patients are considered for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Carboplatin, Vincristine Sulfate, Temozolomide): Induction therapy: Patients receive carboplatin IV (175/m2) over 1 hour on days 1, 8, 15, and 22; vincristine IV (1.5 mg/m2) on days 1, 8, 15, 22, 29, and 36; and oral temozolomide (200 mg/m2) on days 43-47. Four weeks after the completion of induction therapy, patients achieving stable or responding disease proceed to maintenance therapy. Maintenance therapy: Patients receive carboplatin (175/m2) and temozolomide (200 mg/m2) as in induction therapy and vincristine IV ((1.5 mg/m2) day 1 of weeks 10,11,12. Treatment repeats every 10 weeks for a total of 6 courses in the absence of disease progression.
  carboplatin: Given IV
  temozolomide: Given orally
  vincristine sulfate: Given IV
Arm/Group | Carboplatin, Vincristine Sulfate, Temozolomide)
Number analyzed (Participants) | 65
Participants | 0

4. Secondary Outcome: Number of Participants Who Experienced a Grade 3 or 4 Thrombocytopenia and/or Neutropenia.
Description: Occurence of grade 3 or 4 thrombocytopenia or neutropenia while receiving protocol therapy.
Time Frame: Up to 18 months of protocol therapy
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin, Vincristine Sulfate, Temozolomide)
Number analyzed (Participants) | 65
Participants | 43

5. Secondary Outcome: Percent Probability of Progression-free Survival (PFS)
Description: Percentage probability of being alive and without the occurrence of disease progression 3 years following enrollment.
Time Frame: 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percent probability PFS
Arm/Group | Carboplatin, Vincristine Sulfate, Temozolomide)
Number analyzed (Participants) | 65
Percent probability PFS | 60.59 [47.48 to 71.40]

6. Secondary Outcome: Percentage Probability of Event-free Survival (EFS)
Description: Percentage probability of being alive and without the occurrence of disease progression or second malignant neoplasm 6 years following enrollment.
Time Frame: Six years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percent probability EFS
Arm/Group | Carboplatin, Vincristine Sulfate, Temozolomide)
Number analyzed (Participants) | 65
percent probability EFS | 40.89 [28.63 to 52.76]

7. Secondary Outcome: Total Number of Patients Experiencing a Response
Description: Response as complete response, partial response, stable disease, or progressive disease using three-dimensional imaging measurements (preferable) or two-dimensional imaging measurements, as well as the response in the context of multiple lesions or disseminated disease.
Time Frame: Up to 18 months of protocol therapy
Population: Sixty-five (65) eligible patients were enrolled and received protocol therapy. Of these patients, 60 had data submission sufficient to determine response.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin, Vincristine Sulfate, Temozolomide)
Number analyzed (Participants) | 60
Participants
  Complete response | 2
  Partial response | 15
  Stable disease | 36
  Progressive disease | 7

ADVERSE EVENTS:
Description: 66 patients enrolled, 64 reported for adverse events as 1 patient was ineligible and 1 patient missed a reporting period.
Arm/Group | Treatment (Carboplatin, Vincristine Sulfate, Temozolomide)
Serious Adverse Events (participants affected / at risk) | 6/64
Other Adverse Events (participants affected / at risk) | 50/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Carboplatin, Vincristine Sulfate, Temozolomide) (N=64)
Alanine aminotransferase increased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Proteinuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Carboplatin, Vincristine Sulfate, Temozolomide) (N=64)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 10
Acidosis (Metabolism and nutrition disorders) | 10
Agitation (Psychiatric disorders) | 3
Alanine aminotransferase increased (Investigations) | 19
Alkaline phosphatase increased (Investigations) | 7
Allergic reaction (Immune system disorders) | 7
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 10
Anaphylaxis (Immune system disorders) | 7
Anemia (Blood and lymphatic system disorders) | 33
Anorexia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 21
Ataxia (Nervous system disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blood antidiuretic hormone abnormal (Investigations) | 2
Blood bilirubin increased (Investigations) | 3
Blood corticotrophin decreased (Investigations) | 1
Blurred vision (Eye disorders) | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 3
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Catheter related infection (Infections and infestations) | 2
Cholesterol high (Investigations) | 1
Cognitive disturbance (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Creatinine increased (Investigations) | 3
Cushingoid (Endocrine disorders) | 3
Cystitis noninfective (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Diarrhea (Gastrointestinal disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Edema face (General disorders) | 2
Enterocolitis infectious (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Esophageal infection (Infections and infestations) | 1
Extraocular muscle paresis (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 3
Eye infection (Infections and infestations) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 10
Fever (General disorders) | 18
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Gum infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 11
Hydrocephalus (Nervous system disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 23
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 9
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hypoglycemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 14
Hypophosphatemia (Metabolism and nutrition disorders) | 10
Hypotension (Vascular disorders) | 2
Ileus (Gastrointestinal disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 11
Insomnia (Psychiatric disorders) | 2
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 1
Investigations - Other, specify (Investigations) | 1
Irritability (General disorders) | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Lymphocyte count decreased (Investigations) | 17
Memory impairment (Nervous system disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 4
Neutrophil count decreased (Investigations) | 42
Non-cardiac chest pain (General disorders) | 1
Oculomotor nerve disorder (Nervous system disorders) | 2
Optic nerve disorder (Eye disorders) | 1
Oral pain (Gastrointestinal disorders) | 3
Otitis media (Infections and infestations) | 3
Pain (General disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 7
Personality change (Psychiatric disorders) | 3
Pharyngitis (Infections and infestations) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Photophobia (Eye disorders) | 2
Platelet count decreased (Investigations) | 30
Pruritus (Skin and subcutaneous tissue disorders) | 4
Purpura (Skin and subcutaneous tissue disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Rectal hemorrhage (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4
Rhinitis infective (Infections and infestations) | 1
Seizure (Nervous system disorders) | 3
Serum sickness (Immune system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Toothache (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 5
Trigeminal nerve disorder (Nervous system disorders) | 3
Upper respiratory infection (Infections and infestations) | 3
Urinary frequency (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Vaginal inflammation (Reproductive system and breast disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 23
Watering eyes (Eye disorders) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 5
White blood cell decreased (Investigations) | 31
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Wound infection (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No